CLINICAL TRIAL: NCT02609776
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of JNJ-61186372, a Human Bispecific EGFR and cMet Antibody, in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Amivantamab, a Human Bispecific EGFR and cMet Antibody, in Participants With Advanced Non-Small Cell Lung Cancer
Acronym: CHRYSALIS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108064; 61186372EDI1001 (Other: Janssen Research & Development, LLC); 2018-003908-38 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; Amivantamab; First-in-Human; Human Bispecific Epidermal Growth Factor Receptor (EGFR); c-Mesenchymal-Epithelial Transition (cMet) Antibody; JNJ372; Exon 20; Exon 20 insertion; Tyrosine Kinase Inhibitor (TKI) Resistant; TKI Resistance; EGFR C797s; Met Amplification; Met + EGFR bispecific
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; lazertinib; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1:Amivantamab Monotherapy+Combination Dose Escalations (Experimental): The first cohort of participants will receive intravenous (IV) infusions of Amivantamab 140 milligram (mg) as monotherapy. Each subsequent cohort will receive IV infusions of Amivantamab at increased dose level. Dose escalation will continue until maximum tolerated dose is reached or all planned doses are administered. Participants will receive IV infusion of Amivantamab once weekly during cycle 1 and once every 2 weeks during subsequent cycles (duration of each treatment cycle is 28 days). Participants will receive lazertinib and Amivantamab on Cycle 1 Day 1 (C1D1) prior to initiation of Amivantamab (C1D1) at predefined dose levels, based upon observed safety and protocol defined criteria. Lazertinib will be administered daily thereafter, on 28-day Amivantamab treatment cycle. In Chemotherapy Combination Cohort, participants will receive Amivantamab, administered on a 21-day cycle, in combination with standard of care carboplatin and pemetrexed.
  Interventions: Drug: Amivantamab; Drug: Lazertinib; Drug: Carboplatin; Drug: Pemetrexed
- Part 2:Amivantamab Monotherapy+Combination Dose Expansion (Experimental): Participants will receive IV infusion of Amivantamab as monotherapy at Phase 2 dose (RP2D) regimen or in combination lazertinib at the recommended Phase 2 combination dose (RP2CD) regimen as determined in Part 1. The purpose of dose expansion is to further evaluate safety, tolerability, pharmacokinetic, and to assess preliminary efficacy in monotherapy and combination therapy cohorts.
  Interventions: Drug: Amivantamab; Drug: Lazertinib

INTERVENTIONS:
Drug: Amivantamab — The first cohort of participants will receive IV infusions of Amivantamab 140 mg as monotherapy. Each subsequent cohort will receive IV infusions of Amivantamab at increased dose level until maximum tolerated dose is reached or all planned doses are administered. Participants will receive lazertinib and Amivantamab at predefined dose levels, based upon observed safety and protocol defined criteria. The duration of each treatment cycle is 28 days. In Chemotherapy Combination Cohort, participants will receive Amivantamab, administered on a 21-day cycle, in combination with the administration of standard of care carboplatin and pemetrexed.
  Other Names: JNJ-61186372
  Arms: Part 1:Amivantamab Monotherapy+Combination Dose Escalations
Drug: Amivantamab — Participants will receive IV infusion of Amivantamab as monotherapy at RP2D regimen or in combination lazertinib at RP2CD regimen as determined in Part 1.
  Other Names: JNJ-61186372
  Arms: Part 2:Amivantamab Monotherapy+Combination Dose Expansion
Drug: Lazertinib — Lazertinib will be administered in combination with Amivantamab at predefined dose levels, based upon observed safety and protocol defined criteria. Lazertinib will be administered daily on the 28-day Amivantamab treatment cycle.
  Other Names: JNJ-73841937; YH25448
Drug: Carboplatin — Participants will receive carboplatin in combination with pemetrexed and Amivantamab as an IV infusion on 21-day treatment cycle in Part 1 Chemotherapy Combination Cohort only.
  Arms: Part 1:Amivantamab Monotherapy+Combination Dose Escalations
Drug: Pemetrexed — Participants will receive pemetrexed in combination with carboplatin and Amivantamab as an IV infusion on 21-day treatment cycle in Part 1 Chemotherapy Combination Cohort only.
  Arms: Part 1:Amivantamab Monotherapy+Combination Dose Escalations

SUMMARY:
The purpose of study is to evaluate the safety, pharmacokinetics, and preliminary efficacy of Amivantamab as a monotherapy and in combination with lazertinib, and to determine the recommended Phase 2 dose (RP2D) (monotherapy), recommended Phase 2 combination dose (RP2CD) (combination therapy), and to determine recommended Phase 2 Dose (RP2q3W) with combination chemotherapy (Amivantamab in combination with standard of care carboplatin and pemetrexed) in 21 day treatment cycle for participants with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This open label (all participants know the identity of the study drug), multicenter (more than one study site), first-in-human study consists of 2 parts. Part 1 is a Amivantamab Monotherapy and Combination Dose Escalations and Part 2 Amivantamab Monotherapy and Combination Dose Expansions. In Part 1, participants with evaluable NSCLC will be enrolled into cohorts at increasing dose levels of Amivantamab monotherapy, the RP2CD of the Amivantamab and lazertinib combination which will be administered in 28 day treatment cycles, and RP2q3W of Amivantamab in combination with standard of care carboplatin and pemetrexed (chemotherapy combination) which will be administered in 21 day treatment cycles. The dose will be escalated until the maximum tolerated dose (MTD, or maximum administered dose [MAD], if no MTD is found) is reached. Part 1 will follow a traditional 3+3 design. At each dose level, 3 participants will complete Cycle 1. If no dose limiting toxicity (DLT) occurs in these 3 participants, then escalation will continue in a new cohort of 3 participants. Data from Part 1 will be used to determine one or more RP2D regimen(s). In Part 2, participants with documented epidermal growth factor receptor (EGFR) mutations and measurable disease, whose disease has progressed after previous treatment will be enrolled and receive Amivantamab at the RP2D determined in Part 1 as a monotherapy at the RP2D regimen(s), or in combination with lazertinib at the RP2CD regimen. For both parts, the study consists of following periods: an optional pre-Screening period; a Screening period (up to 28 days prior to the first dose of study drug); a Treatment period (first dose of study drug until 30(+7) days after the last dose of study drug or prior to starting any subsequent anti-cancer treatment, whichever comes first); and a Follow Up period (approximately 6 months). All participants will be followed for survival in the post-treatment follow-up period until the end of study and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) that is metastatic or unresectable. Participants must have either progressed after prior standard of care therapy (Cohorts C and hepatocyte growth factor receptor gene [MET]-1: epidermal growth factor receptor [EGFR] tyrosine kinase inhibitor [TKI]; Cohort D: platinum-based chemotherapy; MET-2: per regional standard of care; Cohorts wild-type adenocarcinoma (WT-Ad) and wild-type squamous cell carcinoma (WT-Sq): platinum-containing chemotherapy and programmed death- 1/ ligand-1 (PD-1/L1) therapy, either as a combined regimen or as separate lines of therapy) for metastatic disease, or be ineligible for, or have refused all other currently available therapeutic options. In cases where participants refuse currently available therapeutic options, this must be documented in the study records. For Part 1 Chemotherapy Combination Cohort only: Participants must have histologically or cytologically confirmed NSCLC that is metastatic or unresectable and be eligible for treatment with combination carboplatin and pemetrexed, in accordance with standard of care, and be willing to receive additional investigational therapy with Amivantamab
* For Part 1 Combination Dose Escalation with lazertinib only: Participants must have been diagnosed with EGFR Exon 19del or L858R activating mutation and (a) be treatment naïve for metastatic disease, without access to third generation TKI in the front-line setting, or (b) have progressed after front-line treatment with first (erlotinib or gefitinib) or second generation (afatinib) TKI and are ineligible for Cohort MET-1, or (c) have been treated with a third generation TKI (e.g., osimertinib) in either the front line or second-line setting, and are not eligible for enrollment in either Cohort C or MET-1. For Part 1 Chemotherapy Combination Cohort: Participants may be diagnosed with EGFR mutated or EGFR wild type NSCLC. For Part 2 Cohorts C, D, MET-1, and MET-2 only: Participants must also have disease with a previously diagnosed activating epidermal growth factor receptor (EGFR) mutation (includes both inhibitor sensitive primary mutations such as Exon 19 deletion and L858R (Cohort C, E, and MET-1), as well as marketed TKI-resistant mutations such as Exon 20 insertion (Cohort C, D and MET-1) or activating cMet Exon 14 skipping mutation (Cohort MET-2). Documentation of primary activating EGFR or cMet mutation eligibility by CLIA-certified laboratory (or equivalent) testing is required. For Part 2 Cohorts WT-Ad and WT-Sq: Participants must have wild-type EGFR, anaplastic lymphoma kinase (ALK), and absence of MET Exon 14 skipping mutation as tested by the Food and Drug Administration (FDA) approved test or a CLIA-certified laboratory (or equivalent). The pathology report or equivalent must be in the medical record for verification. Where testing for EGFR and ALK are not part of standard of care for participants with squamous cell carcinoma histology, documentation of the absence of these mutations is not necessary for enrollment into the WT-Sq cohort
* For Part 1: Participant must have evaluable disease. For Part 2: Participant must have measurable disease according to Response Criteria in Solid Tumors (RECIST) v1.1
* For Part 2: Cohorts A and B: Participants EGFR mutated disease must have most recently progressed following treatment with a marketed EGFR inhibitor. Exception: In participants diagnosed with mutations associated with de novo EGFR inhibitor resistance (for example, Exon 20 insertions), only previous treatment with combination platinum-based chemotherapy is required. Cohort C: Participants with primary EGFR mutated disease, with a documented EGFR alteration (example, C797S) mediating resistance to previous treatment with a third generation EGFR TKI (for example, osimertinib), in participants with primary Exon 20ins disease, the documented EGFR alteration may arise following treatment with a TKI with known activity against Exon 20ins disease (for example, poziotinib). Cohort D: participants must have been previously diagnosed with an EGFR Exon 20 insertion and have not been previously treated with a TKI with known activity against Exon 20ins disease (example, poziotinib). Cohort MET-1: Participants with documented primary EGFR mutated disease and documented MET amplification or MET mutation after progression on any EGFR TKI. Participants with disease characterized by both MET amplification and EGFR resistance mutations to prior third generation EGFR TKI will be preferentially enrolled into Cohort C. Participants may have received or have been intolerant to prior platinum-based chemotherapy. Cohort MET-2: Participants with documented primary MET Exon 14 skipping mutation non-small cell lung cancer (NSCLC). Cohort E (combination Amivantamab and lazertinib): Participants must have been diagnosed with EGFR Exon 19del or L858R activating mutation and have progressed after first or second-line treatment with a third generation TKI (e.g., osimertinib). Cohort WT-Ad: Participant must have been diagnosed with NSCLC of adenocarcinoma histology, with positive EGFR and/or MET expression as detected on a validated immunohistochemistry (IHC) assay performed by the central laboratory and have progressed on prior platinum containing chemotherapy and PD-1/L1 therapy, either as a combined regimen or as a separate line of therapy. Eligibility may be determined through IHC analysis of either archival (pre-screening) or mandatory fresh tumor tissue collected during the Screening period. Cohort WT-Sq: Participant must have been diagnosed with NSCLC of squamous cell carcinoma histology, with positive EGFR and/or MET expression as detected on a validated IHC assay performed by the central laboratory and have progressed on prior platinum-containing chemotherapy and PD-1/L1 therapy, either as a combined regimen or as a separate line of therapy. Eligibility may be determined through IHC analysis of either archival (pre-screening) or mandatory fresh tumor tissue collected during the Screening
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Participant has uncontrolled inter-current illness, including but not limited to poorly controlled hypertension, or diabetes, ongoing or active infection, (that is, has discontinued all antibiotics for at least one week prior to first dose of study drug), or psychiatric illness/social situation that would limit compliance with study requirements. Participants with medical conditions requiring chronic continuous oxygen therapy are excluded. For Part 1 Chemotherapy Combination Cohort only: additionally, participants with active bleeding diathesis
* Participant has had prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks or 4 half-lives whichever is longer, before the first administration of study drug. For agents with long half-lives, the maximum required time since last dose is 4 weeks. Toxicities from previous anti-cancer therapies should have resolved to baseline levels or to Grade 1 or less, (except for alopecia [any grade], Grade less than or equal to [<=] 2 peripheral neuropathy, and Grade less than [<] 2 hypothyroidism stable on hormone replacement). For Part 1 Combination Dose Escalation: Any previous treatment with systemic anti-cancer immunotherapy, including but not limited to anti-PD-1, anti-PD-L1, and anti-CTLA-4 agents. For Part 1 Chemotherapy Combination Cohort only: Any previous treatment with systemic anti-cancer immunotherapy in the past 3 months or localized radiotherapy to lung within the past 6 months. For Part 2 only: Cohorts A and B: Prior treatment with chemotherapy for metastatic disease is not allowed unless the tumor mutation carries de-novo resistance to EGFR TKI (example, Exon 20 insertions). Cohort C and MET-1: Prior treatment with more than 2 lines of cytotoxic chemotherapy for metastatic disease (maintenance therapy is not included). Cohort D: Previous treatment with an EGFR TKI with activity against EGFR Exon 20 insertions (such as poziotinib). Cohort E (combination Amivantamab and lazertinib): Any previous treatment in the metastatic setting with other than a first, second, or third generation EGFR TKI. Cohorts WT-Ad and WT-Sq: more than three lines of prior systemic therapy in the metastatic setting
* Participants with untreated brain metastases. Participants with definitively, locally-treated metastases that are clinically stable and asymptomatic for at least 2 weeks and who are off or receiving low-dose corticosteroid treatment (<=10 mg prednisone or equivalent) for at least 2 weeks prior to study treatment are eligible. Exception: participants with asymptomatic, untreated brain metastases, each less than 1 cm in diameter, may be eligible for Amivantamab and lazertinib combination therapy in the Part 1 Combination Dose Escalation or Part 2 Combination Expansion Cohort E
* Participant has a history of malignancy other than the disease under study within 3 years before Screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with or minimal risk of recurrence within a year from Screening)
* Participant has not fully recovered from major surgery or significant traumatic injury prior the first dose of study drug or expects to have major surgery during the study period or within 6 months after the last dose of study drug
* Participant has, or will have, any of the following: a. An invasive operative procedure with entry into a body cavity, within 4 weeks or without complete recovery before Cycle 1 Day 1. Thoracentesis, if needed, and percutaneous biopsy for baseline tumor tissue sample may be done less than 4 weeks prior to Cycle 1 Day 1, as long as the participant has adequately recovered from the procedure prior to the first dose of study drug in the clinical judgement of the investigator; b. Significant traumatic injury within 3 weeks before the start of Cycle 1 Day 1 (all wounds must be fully healed prior to Day 1); c. Any medical condition that requires intact wound healing capacity and is expected to endanger subject safety if wound healing capacity would be severely reduced during administration of the investigational agent; d. Expected major surgery while the investigational agent is being administered or within 6 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose Limiting Toxicity (DLT) | Up to Day 28
  The Dose Limiting Toxicity (DLT) is based on drug related adverse events and includes unacceptable hematologic toxicity, non-hematologic toxicity of Grade 3 or higher, or elevations in hepatic enzymes suggestive of drug-induced liver injury.
Part 2: Number of Participants With Adverse Events (AEs) and Serious AEs | Screening up to follow-up (30 [+7] days after the last dose)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 2: Overall Response Rate (ORR) | Up to End of Treatment Follow (EOT) Up Period (30 [+7] days after the last dose)
  Overall response rate (ORR) is defined as the percentage of participants who achieve either a CR or PR as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). CR: disappearance of all target lesions and non-target lesions. All lymph nodes must be non-pathological in size (< 10 mm short axis) and normalisation of tumour marker levels; PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters and Persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits.
Part 2: Duration of Response (DOR) | Up to EOT Follow Up Period (30 [+7] days after the last dose)
  DOR will be calculated as time from initial response of CR (disappearance of all target lesions and non-target lesions. All lymph nodes must be non-pathological in size ([<] 10 [mm] short axis) and normalisation of tumour marker levels) or PR (at least a 30 [%] decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters and persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits or durable stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study and persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits) to progressive disease (PD) or death due to underlying disease, whichever comes first, only for participants who achieve CR or PR.
Part 2: Percentage of Participants With Clinical Benefit | Up to EOT Follow Up Period (30 [+7] days after the last dose)
  Clinical benefit rate is defined as the percentage of participants achieving complete response (CR): disappearance of all target lesions and non-target lesions. All lymph nodes must be non-pathological in size (less than [<] 10 millimeter [mm] short axis) and normalisation of tumour marker levels or partial response (PR): at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters and persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits or durable stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study and persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits.
Trough Serum Concentration (Ctrough) of Amivantamab | Up to EOT (30 days after last dose)
  Ctrough is the observed serum concentration immediately prior to the next administration.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Amivantamab | Up to EOT (30 days after last dose)
  The AUCtau is the area under the serum concentration-time curve during a dose interval time period (tau)

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Amivantamab | Cycle 1 Day 1: predose through end of infusion (EOT) or Follow Up (approximately 16 months) (each cycle is of 28 days)
  The Cmax is the maximum observed serum concentration of Amivantamab.
Time to Reach Maximum Observed Serum Concentration (Tmax) of Amivantamab | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  The Tmax is defined as time to reach maximum observed serum concentration of Amivantamab.
Area Under the Serum Concentration-Time Curve From t1 to t2 Time (AUC[t1-t2]) of Amivantamab | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  The AUC(t1-t2) is the area under the serum Amivantamab concentration-time curve from time t1 to t2.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Amivantamab | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  The AUCtau is the area under the serum concentration-time curve during a dose interval time period (tau)
Trough Serum Concentration (Ctrough) of Amivantamab | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  The Ctrough is the observed serum concentration immediately prior to the next administration.
Maximum Serum Concentration (Cmax) of Lazertinib | Cycle 1 Day 1: predose through EOT (30 [+7] days after last dose [Cycle 4 Day 15]) (each cycle is of 28 days)
  Cmax is the maximum observed serum concentration of lazertinib.
Time to Reach Maximum Observed Serum Concentration (Tmax) of Lazertinib | Cycle 1 Day 1: predose through EOT (30 [+7] days after last dose [Cycle 4 Day 15]) (each cycle is of 28 days)
  Tmax is defined as time to reach maximum observed serum concentration of lazertinib.
Trough Serum Concentration (Ctrough) of Lazertinib | Cycle 1 Day 1: predose through EOT (30 [+7] days after last dose [Cycle 4 Day 15]) (each cycle is of 28 days)
  Ctrough is the observed serum concentration immediately prior to the next administration.
Accumulation ratio (R) of Amivantamab | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  The R is the accumulation ratio calculated as Cmax or AUC after multiple doses divided by Cmax or AUC after the first dose, respectively.
Number of Participants With Anti-Drug Antibodies (ADA) | Cycle 1 Day 1: predose through EOT or Follow Up (approximately 16 months)
  Serum levels of antibodies to Amivantamab for evaluation of potential immunogenicity.
Progression-Free Survival (PFS) | Up to End of Treatment Follow Up Period (30 [+7] days after the last dose)
  PFS is defined as the time from first infusion of study drug to PD or death due to any cause.
Time to Treatment Failure (TTF) | Up to End of Treatment Follow Up Period (30 [+7] days after the last dose)
  TTF is defined as the time from the first infusion of the study drug to discontinuation of treatment for any reason, including disease progression, treatment toxicity, death, and will be utilized to capture clinical benefit for patients continuing treatment beyond RECIST v1.1 defined disease progression.
Overall Survival (OS) | Up to End of Treatment Follow Up Period (30 [+7] days after the last dose)
  OS is defined as the time from first infusion of study drug to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (69):
- United States (17):
  - Duarte, California
  - La Jolla, California
  - Orange, California
  - Santa Monica, California
  - West Hollywood, California
  - Tampa, Florida
  - Chicago, Illinois
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Fairfax, Virginia
- Australia (5):
  - Camperdown
  - Heidelberg
  - Kogarah
  - Murdoch
  - Woolloongabba
- Toronto, Ontario, Canada
- China (12):
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Hefei
  - Nanchang
  - Nanjing
  - Wuhan
  - Zhengzhou
- France (7):
  - Bordeaux
  - Dijon
  - Lyon
  - Marseille
  - Paris
  - Saint-Herblain
  - Villejuif
- Japan (10):
  - Chūōku
  - Hyōgo
  - Kashiwa
  - Kurume
  - Nagoya
  - Niigata
  - Osaka
  - Tokyo
  - Wakayama
  - Yonago
- South Korea (5):
  - Cheongju-si
  - Goyang-si
  - Incheon
  - Seongnam-si
  - Seoul
- Spain (6):
  - A Coruña
  - Barcelona
  - Madrid
  - Málaga
  - Santander
  - Seville
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (3):
  - Manchester
  - Newcastle upon Tyne
  - Sutton

REFERENCES:
- [Derived] Lenz G, Pereira RA, Schwengber WK, Tumelero M, Peruzzo N, Lago LS, Lopes G. Premature Deaths and Life-Years Lost From Lack of Amivantamab in Brazil's Unified Health System. JCO Glob Oncol. 2025 Nov;11:e2500302. doi: 10.1200/GO-25-00302. Epub 2025 Nov 19. PMID 41259729
- [Derived] Cho BC, Kim DW, Spira AI, Gomez JE, Haura EB, Kim SW, Sanborn RE, Cho EK, Lee KH, Minchom A, Lee JS, Han JY, Nagasaka M, Sabari JK, Ou SI, Lorenzini P, Bauml JM, Curtin JC, Roshak A, Gao G, Xie J, Thayu M, Knoblauch RE, Park K. Amivantamab plus lazertinib in osimertinib-relapsed EGFR-mutant advanced non-small cell lung cancer: a phase 1 trial. Nat Med. 2023 Oct;29(10):2577-2585. doi: 10.1038/s41591-023-02554-7. Epub 2023 Sep 14. PMID 37710001
- [Derived] Spira A, Girard N, Krebs M, Park K, Shu C, Dougherty L, Cho BC. A plain language summary of the results from the group of patients in the CHRYSALIS study with EGFR exon 20 insertion-mutated non-small-cell lung cancer who received amivantamab. Future Oncol. 2023 Oct;19(33):2213-2225. doi: 10.2217/fon-2023-0284. Epub 2023 Aug 17. PMID 37589131
- [Derived] Chon K, Larkins E, Chatterjee S, Mishra-Kalyani PS, Aungst S, Wearne E, Subramaniam S, Li Y, Liu J, Sun J, Charlab R, Zhao H, Saritas-Yildirim B, Bikkavilli RK, Ghosh S, Philip R, Beaver JA, Singh H. FDA Approval Summary: Amivantamab for the Treatment of Patients with Non-Small Cell Lung Cancer with EGFR Exon 20 Insertion Mutations. Clin Cancer Res. 2023 Sep 1;29(17):3262-3266. doi: 10.1158/1078-0432.CCR-22-3713. PMID 37022784
- [Derived] Chouaid C, Bosquet L, Girard N, Kron A, Scheffler M, Griesinger F, Sebastian M, Trigo J, Viteri S, Knott C, Rodrigues B, Rahhali N, Cabrieto J, Diels J, Perualila NJ, Schioppa CA, Sermon J, Toueg R, Erdmann N, Mielke J, Nematian-Samani M, Martin-Fernandez C, Pfaira I, Li T, Mahadevia P, Wolf J. An Adjusted Treatment Comparison Comparing Amivantamab Versus Real-World Clinical Practice in Europe and the United States for Patients with Advanced Non-Small Cell Lung Cancer with Activating Epidermal Growth Factor Receptor Exon 20 Insertion Mutations. Adv Ther. 2023 Mar;40(3):1187-1203. doi: 10.1007/s12325-022-02408-7. Epub 2023 Jan 18. PMID 36652175
- [Derived] Jatkoe T, Wang S, Odegaard JI, Velasco Roth AM, Osgood D, Martinez G, Lucas P, Curtin JC, Karkera J. Clinical Validation of Companion Diagnostics for the Selection of Patients with Non-Small Cell Lung Cancer Tumors Harboring Epidermal Growth Factor Receptor Exon 20 Insertion Mutations for Treatment with Amivantamab. J Mol Diagn. 2022 Nov;24(11):1181-1188. doi: 10.1016/j.jmoldx.2022.07.003. Epub 2022 Aug 10. PMID 35963523
- [Derived] Park K, Haura EB, Leighl NB, Mitchell P, Shu CA, Girard N, Viteri S, Han JY, Kim SW, Lee CK, Sabari JK, Spira AI, Yang TY, Kim DW, Lee KH, Sanborn RE, Trigo J, Goto K, Lee JS, Yang JC, Govindan R, Bauml JM, Garrido P, Krebs MG, Reckamp KL, Xie J, Curtin JC, Haddish-Berhane N, Roshak A, Millington D, Lorenzini P, Thayu M, Knoblauch RE, Cho BC. Amivantamab in EGFR Exon 20 Insertion-Mutated Non-Small-Cell Lung Cancer Progressing on Platinum Chemotherapy: Initial Results From the CHRYSALIS Phase I Study. J Clin Oncol. 2021 Oct 20;39(30):3391-3402. doi: 10.1200/JCO.21.00662. Epub 2021 Aug 2. PMID 34339292
- [Derived] Kohler J, Janne PA. Amivantamab: Treating EGFR Exon 20-Mutant Cancers With Bispecific Antibody-Mediated Receptor Degradation. J Clin Oncol. 2021 Oct 20;39(30):3403-3406. doi: 10.1200/JCO.21.01494. Epub 2021 Aug 2. No abstract available. PMID 34339261